CLINICAL TRIAL: NCT02409589
Title: A Randomized Open-labeled Multicenter Study to Assess a New Intracavitary Electrocardiographic Guiding Method for Real-time Positioning the Tip of Three-way Valve Type Peripherally Inserted Central Catheters (PROJECT_EGG)
Brief Title: An Intracavitary Electrocardiographic System for Real-time Positioning Peripherally Inserted Central Catheter Tip
Acronym: PROJECT_EGG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuan Ling (Other)
Responsible Party: Sponsor-Investigator, Yuan Ling, Associate Chief Nurse, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-001
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Peripherally Inserted Central Catheter; Intracavitary Electrocardiogram Guiding
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ECG-guided PICC Tip Placement (Experimental): New intracavitary ECG guiding method
  Interventions: Device: ECG
- Conventional (Active Comparator): Surface prediction length method
  Interventions: Procedure: Surface prediction length method

INTERVENTIONS:
Device: ECG — The ECG-guided PICC tip detection method will be used to identify catheter tip location during the procedural placement of the catheter. This method involves an ECG monitor which will be connected to the guidewire used for catheter placement. The changes in the ECG p-wave will guide correct PICC placement. An X-ray radiograph will be conducted to confirm the tip location after PICC placement.
  Arms: ECG-guided PICC Tip Placement
Procedure: Surface prediction length method — The method will estimate the length of the catheter from puncture site to the junction of superior vena cava / right atrium (SVC-RA) . Tip location is placed according to the estimated length but later on will be determinated by chest X-ray performed after the placement procedure. If the tip location is not at an ideal place, additional procedures and X-ray radiograph would be required in order to ensure proper tip location.
  Arms: Conventional

SUMMARY:
The purpose of this study is to compare a new intracavitary ECG guiding method for real-time positioning the tip of three-way valve type peripherally inserted central catheters versus conventional surface prediction length method in terms of single-time target rate.

DETAILED DESCRIPTION:
The use of peripherally inserted central catheters (PICCs) has increased significantly for cancer patients receiving chemotherapy. For these patients, PICCs afford many advantages with regards to complications and treatment convenience.

Current practice utilizes the estimated length of the catheter from puncture site to the junction of superior vena cava / right atrium (SVC-RA) for guiding tip placement. Next the catheter tip placement was confirmed by radiographic imaging prior to use of the line for administration of chemotherapy medications. In this case, the catheter is often mal-positioned and requires adjustment and repeat radiographic imaging in order to ensure proper placement, ideally at the SVC-RA junction. These potentially additional procedures are time-consuming and also expose patients, nurses and physicians to radiations.

Intracavitary electrocardiogram with an electrode placed inside the catheter during insertion has shown identifiable changes in P-wave, which are sufficient to guide PICC tip placement. Moreover, less procedural time and radiation are expected.

This study aims to demonstrate if this intracavitary electrocardiogram guided method is superior to conventional surface prediction length method in terms of single-time target rate of correct tip placement. In addition, we would like to investigate symptomatic thrombosis incidence and its risk factors after three-valve PICC implanted among patients with malignant tumors; to clarify procedure time used and cost of the new intracavitary ECG guiding method and to explore the maximal P-wave amplitude of intracavity ECG real-time positioning technology and its predictive factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malignant tumors who will require periodical infusion of chemotherapy drugs using three-valve PICC;
2. Aged >18 to < 80 years old;
3. Baseline ECG records prior to PICC catheter showed normal P wave;
4. Agreed to participate in this study, and signed PICC informed consent.

   Exclusion Criteria:
5. Patients with heart diseases, such as valvular heart disease, atrial fibrillation, supraventricular tachycardia, pulmonary heart disease or having a pacemaker and post cardiac surgery which may affect P waves.
6. Patients unable to lie in the prostrate or semi-supine position.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Single-time target rate | Less than 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ling Yuan, Master, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (8):
- China (8):
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - Nanjing Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - The 2nd Affliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - People's Hospital Affiliated to Jiangsu University, Zhenjiang, Jiangsu

REFERENCES:
- [Derived] Yuan L, Li R, Meng A, Feng Y, Wu X, Yang Y, Chen P, Qiu Z, Qi J, Chen C, Wei J, Qin M, Kong W, Chen X, Xu W. Superior success rate of intracavitary electrocardiogram guidance for peripherally inserted central catheter placement in patients with cancer: A randomized open-label controlled multicenter study. PLoS One. 2017 Mar 9;12(3):e0171630. doi: 10.1371/journal.pone.0171630. eCollection 2017. PMID 28278167